CLINICAL TRIAL: NCT06718010
Title: Age-Related Peripheral Blood Components and Their Association With Treatment Efficacy in Breast Cancer Patients: An Observational Cohort Study
Brief Title: The Association Between Age-related Peripheral Blood Components and Treatment Efficacy in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Other Study IDs: ALPHABET-001
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Age
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood sample and tumor sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention (observational study) — The study respects the investigator's choice of treatment, without specifying which drugs should be used, the dosage, the administration mode (including monotherapy, combination therapy, or sequential therapy), or the duration of treatment.

SUMMARY:
This study is a single-center, prospective/retrospective, observational clinical research designed to compare the differences in peripheral blood components between young and elderly HR+HER2- breast cancer patients, and to identify peripheral blood components that may affect the prognosis of young HR+HER2- breast cancer patients.

The study population consists of early-stage HR+HER2- breast cancer patients receiving neoadjuvant therapy. Eligible patients who require neoadjuvant treatment will be enrolled in the study. Retrospective data and samples will be collected based on existing patient medical records and tissue biobank samples. Prospective data collection will be based on routine clinical treatment during the study period and will continue until the patient completes neoadjuvant therapy and undergoes primary tumor surgery, or until the study is prematurely terminated.

HR+HER2- breast cancer patients receiving neoadjuvant therapy will be divided into young and elderly groups. Peripheral blood samples will be collected at baseline (T0, prior to treatment) and after two cycles of neoadjuvant therapy (T1). Paired baseline tumor biopsy samples and/or surgical tumor samples will also be collected. Peripheral blood and tumor samples will undergo appropriate tests.

The study respects the investigator's choice of treatment, without specifying which drugs should be used, the dosage, the administration mode (including monotherapy, combination therapy, or sequential therapy), or the duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent according to local regulations;
2. Age ≥ 18 years;
3. Female;
4. Histologically/cytologically confirmed breast cancer;
5. Determined by immunohistochemistry to be ER+ or PR+ (with at least 1% of cells expressing estrogen receptors) and HER2-.

Exclusion Criteria:

1. Presence of distant metastasis;
2. History of other malignancies. Patients with basal cell carcinoma or squamous cell carcinoma of the skin, cervical carcinoma in situ, or other cancers who have been disease-free for more than 5 years after appropriate treatment may be included;
3. Participation in another clinical trial within 30 days prior to starting neoadjuvant treatment for breast cancer, and receiving investigational drugs or any concomitant treatment including investigational drugs;
4. Immunodeficiency or HIV infection;
5. Severe heart, lung, liver, or kidney dysfunction;
6. Uncontrolled infections or active infections;
7. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of early-stage luminal breast cancer patients receiving neoadjuvant therapy.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood components related to efficacy | Approximately 18 months
  Compare the differences in peripheral blood components between patients with different treatment efficacies.

SECONDARY OUTCOMES:
Age-related components associated with efficacy | Approximately 18 months
  Identify age-related peripheral blood and tissue components associated with efficacy.
Age-related peripheral blood components | Approximately 18 months
  Evaluate the differences in peripheral blood components between young and elderly patients.
Efficacy of neoadjuvant immunotherapy in young and elderly patients assessed by Miller-Payne grading | Approximately 18 months
  Compare the efficacy of neoadjuvant immunotherapy in young and elderly patients assessed by Miller-Payne grading. The Miller-Payne grading system is primarily used to evaluate the efficacy of neoadjuvant therapy in breast cancer. Based on the percentage of residual tumor cells, it is divided into five grades, ranging from Grade I to Grade V, with higher grades indicating a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center Shanghai, China, 200032, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided